CLINICAL TRIAL: NCT05711407
Title: The Relationship of Peri-implantitis With COX-2 Gene Polymorphisms, Active MMP-8 Levels, and Characterization of Associated Microbiota.
Brief Title: Peri-implantitis and MMP-8
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Ioannis Fragkioudakis, PhD Student, Aristotle University Of Thessaloniki
Other Study IDs: Frag3
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Peri-implantitis: Group Case
  Interventions: Genetic: Gene Polymorphisms of MMP-8
- Healthy: Group Control
  Interventions: Genetic: Gene Polymorphisms of MMP-8

INTERVENTIONS:
Genetic: Gene Polymorphisms of MMP-8 — Saliva Samples

SUMMARY:
Peri-implantitis is defined as the pathological condition around dental implants characterized by inflammation in the peri-implant mucosa and progressive bone loss, eventually leading to implant loss. Peri-implantitis is thought to be a disease analogous to periodontitis with a prevalence reaching 22%. Though peri-implantitis is readily recognized as a part of modern dentistry, the exact etiology or an effective treatment regimen hasn't been established yet. Thus, contemporary research is orientating toward acknowledging the aetiologic and risk factors of the disease and of course establishing prognostic markers for disease prevention. Microbiota residing in the subgingival plaque are considered the main etiologic factor of the disease, however, current literature has not concluded on the exact microbial composition of peri-implant lesions. In addition, genetic predisposition has been recognized as a risk factor for disease initiation and progression and several observational studies have addressed the potential association between various gene polymorphisms and the occurrence of peri-implantitis. Lastly, to establish effective preventive measures, several biomarkers have been evaluated as potential diagnostic and prognostic markers of disease progression.

Objectives:

1. To identify the relationship of peri-implantitis with Cycloxygenase-2 (COX-2) and MMP-8 gene polymorphisms. Cyclooxygenase catalyzes the production of prostaglandins (PGs) which are an important inflammatory mediator participating in the pathogenesis of peri-implantitis. In addition, PGE2 expression in the peri-implant crevicular fluid will be assessed.
2. To characterize the microbiota associated with peri-implantitis lesions, using novel identification techniques enabling the identification of specific opportunistic bacteria associated with the disease.
3. To test the diagnostic accuracy of a modern chairside test, using metalloproteinase-8 (MMP-8), an enzyme implicated in the pathogenesis of the disease, as a biomarker of disease progression.

DETAILED DESCRIPTION:
Dental implants have become an integrated part of modern dentistry during the last decades. Since osseointegration (the process of an implant being incorporated into the jawbone) was discovered, implant dentistry has gone substantial steps over time. Dental implants comprise of an endosteal part made of titanium and an external prosthetic part, aiding in the rehabilitation of edentulous patients. They offer the possibility to patients missing one or several teeth to achieve the maximum functional and esthetic results, refraining from traditional dentures that are quite unpleasant. Implant industry is gradually growing. Overall, the global market of dental implants was valued at US$ 2,91 billion in 2016 with more than 8.809 million implants placed annually in the US (1). However, the prevalence of biological complications regarding dental implant supported restorations is growing in the same rate (1).

The term "Peri-implantitis" was introduced in the 1st European Workshop of Periodontology in 1994 and since then numerous definitions have been proposed to describe the bone loss that characterizes the aftermath of implant installation (2,3). Peri-implantitis and peri-implant mucositis are covered under the term peri-implant diseases and are considered analogous to periodontal diseases (4). Currently, peri-implantitis is defined as the pathological condition around dental implants characterized by inflammation in the peri-implant mucosa and progressive bone loss, eventually jeopardizing the fate of the implant (5). The number of studies referring to peri-implantitis have risen in the last 30 years according to PubMed, from 86 papers in the 90s' to a total of 1938 manuscripts until now (1). The prevalence of peri-implantitis is also exhibiting growing rates. In a systematic review, Zitzman and Berglundh in 2008 reported a prevalence ranging from 12 to 56% (3). More recent studies reveal a prevalence of 22% (1-47%) (6), 20% (7), 26% (8), and 28% (9). It should be pointed that in the previous studies the exact prevalence of the disease is difficult to estimate and is dependent on several factors including the diagnostic criteria of the disease and the time point chosen for the evaluation (10). However, it is obvious that peri-implantitis is a growing problem affecting implant dentistry and will certainly be the topic of many future studies.

Several protocols have been proposed for the treatment of peri-implantitis including, non-surgical protocols, with implant decontaminating devices and lasers and surgical protocols such as the use of regenerative materials (11,12) . However, if peri-implantitis is already established, the proposed strategies and recommendations for its treatment can still be considered as empirical. From the existing evidence it seems that nonsurgical therapy is not effective, at least not in advanced cases. Surgical techniques may be necessary to provide us with adequate access to degranulate the inflamed tissues effectively as well as to decontaminate the implant surface (13).

The Consensus report of Workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions concluded that peri-implantitis is an inflammatory process of a microbial origin that causes bone loss (4). In addition, several risk factors have been proposed as potential co-drivers in this entity, including history of periodontitis, smoking, diabetes and poor plaque control (5). Factors such as genetic predisposition and release of titanium particles have also been indicated as potential risk factors (14). The microbial involvement in peri-implantitis initiation and progression has been established, however recent studies suggest that peri-implantitis may be a result of a foreign body reaction, emphasizing the role of the host response in the disease initiation. (15). In other words, the aetiology of the disease is yet to be elucidated. However, using conventional DNA probe and cultural analyses, common periodontopathogenic bacteria have been isolated at both healthy and diseased implant sites (16) and the distribution of the detected species did not markedly differ by clinical implant status (17). However, when compared with healthy implant sites alone, peri-implantitis was associated with higher counts of bacterial species considered as consensus periodontal pathogens including Porphyromonas gingivalis and Tannerella forsythia (18). Moreover, observational studies have indicated that peri-implantitis was more frequently linked with opportunistic pathogens such as Pseudomonas aeruginosa and Staphylococcus aureus ,(19,20) fungal organisms (e.g. Candida albicans, Candida boidinii, Penicillum spp., Rhadotorula laryngis, Paelicomyces spp.),(21,22) and viruses (i.e. human cytomegalovirus, Epstein-Barr virus), (23) thus pointing to a rather complex and heterogenous infection. Therefore, the recognition of the exact bacterial composition of peri-implant lesions is of paramount importance.

A significant observation about implant failures is that usually, a small number of patients lose many implants. This clusterization phenomenon has been identified in many studies (24,25). Weyant and his colleagues examined the survival rate of implants in 598 patients and noticed that more than half of the cases that received multiple implants had more than one failure. They estimated that patients who had one implant lost were 1.3 more likely to lose more implants (26). These findings led to the hypothesis that host factors affect implant survival and therefore genetic predisposition may play an important role in the development of peri-implantitis. Many gene polymorphisms have been evaluated. Initially, most of the studies referred to polymorphisms of cytokines which play a key role in the immune response (27-29), such as the interleukins IL-1α, IL-1β, and their antagonist protein IL-1ra, IL-6, IL-10, IL-17, TNF-α and Transforming Growth Factor-β1 (TGF-β1). Apart from these, various other genes have been investigated, e.g. genes encoding CD14, receptor activator of nuclear factor kappa B ligand (RANKL), microRNAs, bone morphogenetic proteins (BMPs), fibroblast growth factor (FGF), TRAF family member-associated NF-kappa-β activator (TANK), serine/threonine-protein kinase B-Raf (BRAF), calcitonin receptor (CTR), haptoglobin. There are many discrepancies in the results of the above-mentioned studies. Some succeeded to detect possible associations and others not. A more novel gene polymorphism mentioned in genetic studies is that of the cyclooxygenase-2 (COX-2). A single nucleotide polymorphism of COX-2 has been shown to alter the expression of the COX-2 gene. Several studies have found an association among COX-2 gene polymorphisms and periodontitis (30-32). However, in the case of peri-implantitis data is scarce.

The diagnosis of peri-implantitis is based on traditional clinical indices, similar to assessment of periodontal disease. In specific, the diagnosis is established by the presence of bleeding and/or suppuration on gentle probing, increased probing depth compared to previous clinical examinations and the presence of bone loss beyond crestal bone level changes resulting from initial bone remodeling (4). However, recent studies question the diagnostic accuracy of clinical indices as such, supporting that the diagnosis of the disease is far more complex (33). In these regards, novel diagnostic methods have been utilized in order to achieve an early and proper diagnosis of the disease (34). A biomarker, or biological marker is a measurable indicator of some biological state or condition. Biomarkers are often measured and evaluated to examine normal biological processes, pathogenic processes, or pharmacologic responses to a therapeutic intervention, and are useful in the diagnosis and prognosis of a disease. In the case of peri-implantitis several biological molecules have been evaluated as potential biomarkers aiding the diagnosis of the disease. Molecules such as TNF-a, IL-1, RANKL have been associated with peri-implantitis in a variety of studies (34). Lately, matrix metalloproteinase 8, (MMP-8),especially in its active form (aMMP-8) has gained much attention of becoming promising biomarker candidate for diagnosing and assessing the progression and course of these episodic oral inflammatory tissue destructive and degenerative diseases (35,36).

Taken all together, peri-implantitis is a complicated disease with a high prevalence among the population. In addition, current data on the etiology and diagnosis of the disease is controversial.

PROPOSAL OBJECTIVES, STATE OF THE ART AND CHALLENGES

1. To address the relationship of peri-implantitis with COX-2 gene polymorphisms, as there are no similar studies in the literature.
2. To identify the pathogenic microbiota that is associated with the disease using novel bacterial identification methods.
3. To evaluate the diagnostic accuracy of an aMMP-8 Point-of-care chair-side test in peri-implantitis.

The rationale in studying each of the studied objectives will be analyzed in a separate section.

- COX-2 gene polymorphisms. The genetic predisposition is considered a potential risk factor for peri-implantitis as already mentioned. A single nucleotide polymorphism (SNP) is single nucleotide variation at a specific position of the genome. Each variation appears in some appreciable degree within a population. SNPs may occur within coding and non-coding sequences of genes, or in the intergenic regions. Considering degeneracy of the genetic code, SNP within a coding sequence may change the amino acid sequence of the coding polypeptide (nonsynonymous SNP), or not affect the protein sequence (synonymous SNP). SNPs outside protein-coding regions may still regulate gene expression through affecting the transcription factor binding, gene splicing, mRNA degradation, or the sequence of noncoding RNA. Therefore, SNPs underlie differences in our susceptibility to disease. SNPs of inflammatory cytokine genes may affect their expression levels or amino acid sequence and, consequently, the host inflammatory response.

COX-2 converts arachidonic acid into prostaglandin H2, which is the precursor of prostaglandin E2. Prostaglandin E2, which mediates proinflammatory and anti-inflammatory reactions in many tissues (37), is also partly responsible for the activating processes involved in resorption of the alveolar bone during the pathogenesis of periodontitis. Associations of the cyclooxygenase 2(COX-2) gene with periodontitis were first identified in Taiwanese and Chinese case-control populations (30,31) and subsequently validated in a northwest European population. Studies as such involving the COX-2 gene have not been conducted in the case of peri-implantitis yet. However, recent gene expression studied have revealed an increased activity of the COX-2 pathway in the case of peri-implantitis (38,39), implying that COX-2 may play an important role in the pathogenesis of peri-implantitis. The association of peri-implantitis with certain gene polymorphisms will allow for a better understanding of the disease, leading to more effective preventing and treatment strategies.

* Microbial factors associated with peri-implantitis Current data confirm that peri-implant infections are dominated by Gram negative bacteria, similar to periodontal infections, but some cases may harbor a distinct microbiota (20,40,41). Although early reports showed similarities between the peri-implant and periodontal flora, later studies demonstrated that peri-implantitis lesions may present not only consensus periodontal pathogens but also opportunistic microorganisms, such as S.aureus, S. anaerobius, Escherichia coli, Candida and Streptococci spp (18). Furthermore, sequencing methods have also revealed other non-cultivable microorganisms associated with peri-implant disease. Asaccharolytic anaerobic gram-positive rods (AAGPR) such as Eubacterium nodatum, Eubacterium brachy, Slackia exigua, Gemella sanguinis and anaerobic Gram-negative rods (OGNR) like Mitsuokella sp., Treponema lecithinolyticum have been identified (42). The discrepancies among these studies may arise from the different methods used for microbiological sampling and processing (43). The microbiological profile of peri-implant diseases remains an issue of interest and many investigations and reviews have been conducted in order to conclude whether the microbiota is different from that of periodontitis; however, controversies still exist. The latest of the studies conclude that there is insufficient evidence to support the distinct microbiota between peri-implant and periodontal diseases (44,45) whereas others state that they may be different entities in terms of microbiological profile (43). Therefore, further studies need to be conducted, in order to define the microbiological profile of peri-implant tissues. Newest technologies, such as shotgun sequencing of the whole genome of bacteria involved in peri-implantitis would be very useful for this purpose, but no such research has been published up to now. Thus, in this study Next Generation Sequencing will be used will be utilized in order to identify the most purulent microbiota associated with the disease. 16s rRNA sequencing will enable the characterization of the whole taxonomic identity of the peri-implant lesions.
* Diagnostic accuracy of ImplantSafe MMP-8 Biomarker Test. Neutrophil collagenase, also called matrix metalloproteinase (MMP)-8, polymorphonuclear (PMN) leukocyte collagenase, or collagenase-2, has been identified and characterized as a major collagenolytic enzyme that causes active periodontal and peri-implant degeneration (APD) in periodontitis and peri-implantitis (46,47). MMP-8 can resolve and regulate inflammatory and immunological cascades by processing nonmatrix bioactive substrates such as chemokines, cytokines, serpins, and complement components. Physiological levels of MMP-8 can exert protective and defensive anti-inflammatory characteristics (48). Increased levels of especially active MMP-8 (aMMP-8), but not the latent, inactive proform, have been found in periodontitis- and peri-implantitis-affected oral fluids (saliva, mouth rinse, gingival crevicular fluid (GCF), and peri-implant sulcular fluid (PISF)) (49). A key characteristic of active periodontal and peri-implant diseases is the sustained pathological elevation and activation of aMMP-8 in periodontal and peri-implant tissues, which are reflected in oral fluids (50). Consequently, aMMP-8 is a promising biomarker candidate for diagnosing and assessing the progression and course of these episodic oral inflammatory tissue destructive and degenerative diseases (46). More importantly, aMMP-8 in oral fluids can also serve as a predictive and preventive adjunctive biotechnological tool to indicate (49,50) preventive interventions (secondary prevention or supportive periodontal/peri-implant therapy (51,52) and to inhibit or reduce the conversion of gingivitis and mucositis to periodontitis and peri-implantitis, respectively.

Recently, lateral-flow point-of-care (PoC)/chair-side tests (PerioSafe and ImplantSafe), discovered in Finland and further developed in Germany (53), have been developed based on earlier described technologies and monoclonal antibodies (53,54). The tests, PerioSafe and ImplantSafe, and reader (ORALyser) have been developed and manufactured by Medix Biochemica Ltd (Espoo, Finland) and Dentognostics GmbH (Jena, Germany) and are commercially available from Dentognostics GmbH (Jena, Germany). In fact, the PoC/chair-side aMMP-8 lateral-flow immunotests resemble the classical pregnancy and/or recently described HIV-PoC tests (55). The aMMP-8 oral fluid tests can be used according to the manufacturer's instructions (47). PerioSafe measures and analyses the levels of aMMP-8 in mouth rinse and ImplantSafe in PISF and GCF; thus, PerioSafe is patient-specific and ImplantSafe is site-specific (47,53). PerioSafe and ImplantSafe test-sticks can be quantitated by the ORALyser reader in 5 min PoC/chair-side. PerioSafe and ImplantSafe with ORALyser quantitation are reliable, quantitative, noninvasive, safe, and inexpensive adjunctive point-of-care diagnostic tools for diagnosis, screening, monitoring, and prevention of periodontal and peri-implant diseases (47). A pilot case-control peri-implantitis study shows both 100% sensitivity and specificity for ImplantSafe test (56).

Methodology and Implementation:

To achieve the previous aims a case control study has been designed and will be carried on in the department of Periodontology and Implant Biology, Dental School, Aristotle university of Thessaloniki.

A study sample of minimum 100 patients attending the Postgraduate Clinic of Periodontology and Implant Biology of Dental School Aristotle University of Thessaloniki for periodontal or peri-implant treatment, will be recruited. Patients should be diagnosed with peri-implantitis according the latest (2017)(4) criteria. The study protocol will be applied to the Ethical Committee of the Faculty of Dentistry of the Aristotle University of Thessaloniki for approval and all patients will be asked to sign their inform consent.

- Work Packages: i. COX-2 gene polymorphisms: Buccal swab will be obtained from all the patients included in the study. After DNA extraction, a polymerase chain reaction (PCR) process will be performed in order to identify the proposed polymorphisms, using commercial primers specific for the gene. The gene polymorphism analyses, and relevant laboratory process will be carried out with the collaboration of the school of Biology, Faculty of Sciences, Aristotle University of Thessaloniki. More specifically, the samples will be collected from Ioannis Fragkioudakis (Postgraduate student of the Department of Periodontology and Implant Biology, Department of Dentistry, Aristotle University of Thessaloniki) and will be stored in -80°C until further processing. The samples will be analyzed in cooperation with the department of Biology, Aristotle university of Thessaloniki under supervision of Professor Minas Arsenakis. The process will be carried out by Ioannis Fragkioudakis and the PhD candidate Symela Koutounidou. The selection of this collaborating organism is based on the previous experience of Professor Minas Arsenakis in gene polymorphisms analysis and the fully equipped laboratory located in the department of Biology AUTh. In addition, the PI, declares successful previous collaborations with the members of the selected organization.

ii. Pathogenic Microbiota Samples will be obtained from the selected implants by the insertion of sterile endodontic paper points into each peri-implant crevice. More specifically, the samples will be collected from Ioannis Fragkioudakis (Postgraduate student of the Department of Periodontology and Implant Biology, Department of Dentistry, Aristotle University of Thessaloniki) and will be stored in -80°C until further processing The samples will be analyzed using Next Generation Sequencing (NGS). More specifically ,16S rRNA sequencing and HOMINGS will be used to identify the whole microbiota included in the samples, enabling the characterization of all the taxonomic levels of bacteria. The NGS will be conducted in collaboration with the department of microbiology, Medical School, A.U.Th. The choice of the collaborating organism and members is based on the availability on the needed laboratory equipment (Access provides by the associated professor Lemonia Skoura) in the AHEPA university general Hospital of Thessaloniki. In addition, the needed laboratory work will be conducted by Fani Chatzopoulou (PhD Student), familiar with the processes, under the supervision of the Associate Professor Dimitrios Chatzidimitriou.

iii. MMP-8 Analysis ImplantSafe rapid aMMP8 analysis tests will be used for the evaluation of the MMP-8 levels in the selected implants. The process will be as follows: Matrix metalloproteinase (MMP)-8 (neutrophil collagenase-2) levels in its active form (aMMP-8) will be collected from the Peri-implant Crevicular Fluid, with the aid of the paper strips included in the test. Afterwards the samples will be analyzed quantitatively by the digital reader ORALyzer® according to the manusfacturer's instructions giving an instant quantification of the aMMP-8 levels. The ORALyzer has been in the possession of the Department of Periodontology since 2019. All the samples will be collected and analyzed by Ioannis Fragkioudakis.

ELIGIBILITY:
Inclusion:

* Screw Retained implant restorations
* Loaded for > 12 months
* Patients Treated for Periodontal Disease

Exclusion

* 3 months patients should have not received antibiotics
* Diabetes and immunosuppressant diseases
* Periodontal maintenance in the previous 3 months

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A study sample of minimum 100 patients attending the Postgraduate Clinic of Periodontology and Implant Biology of Dental School Aristotle University of Thessaloniki for periodontal or peri-implant treatment, will be recruited. Patients should be diagnosed with peri-implantitis according the latest (2017)(4) criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Gene polymorphisms of MMP-8 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dimitra Sakellari, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle Un, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No